CLINICAL TRIAL: NCT01231841
Title: Protocol for Prospective Phase II Study of Rabbit Antithymocyte Globulin (r-ATG/Thymoglobulin) and Cyclosporine (CsA) as a First Line Immunosuppressive (IS) Therapy for Severe Aplastic Anemia (sAA)
Brief Title: Anti-thymocyte Globulin and Cyclosporine as First-Line Therapy in Treating Patients With Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF7922; NCI-2010-01365 (Other: NCI/CTRP)
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Results first posted 2012-03-09 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2018-01

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclosporine; Cyclosporins; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rATG + Cyclosporine (Experimental): Patients receive anti-thymocyte globulin IV daily over 4-24 hours on days 1-5. Beginning on day 6, patients receive oral cyclosporine twice daily for 6 months followed by a taper. Treatment continues in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: cyclosporine; Biological: anti-thymocyte globulin

INTERVENTIONS:
Drug: cyclosporine — Given orally
  Other Names: 27-400; ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin

SUMMARY:
RATIONALE: Immunosuppressive therapies, such as anti-thymocyte globulin and cyclosporine, may improve bone marrow function and increase blood cell counts. PURPOSE: This phase II trial is studying how well giving anti-thymocyte globulin together with cyclosporine as first-line therapy works in treating patients with severe aplastic anemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: To determine the response rate of r-ATG and CsA in the first line setting. SECONDARY OBJECTIVES: To determine the level of IS as assessed by Immuknow assay in responders and compare it to non-responders. OUTLINE:Patients receive anti-thymocyte globulin IV over 4-24 hours daily on days 1-5. Beginning on day 6, patients receive oral cyclosporine twice daily for 6 months followed by a taper. Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* All patients with sAA as defined by Camitta who are candidates for IS therapy; these criteria include bone marrow cellularity < 25% or 25-50% with < 30% of hematopoietic cells; it should also have two of the following three parameters: peripheral blood neutrophils < 0.5 x 10^9/L, platelets < 20 x 10^9/L and reticulocytes < 60 x 10^9/L in anemic patients
* If cytogenetic testing has been done, it should show normal karyotype or be not informative
* Patients should be either unwilling or otherwise ineligible (age, comorbidities, lack of donor) for bone marrow transplantation as a therapeutic modality
* Not previously treated with ATG for sAA
* Patients must have ECOG performance status of 0, 1, or 2
* Vitamin B12 and folic acid deficiency must be ruled out by measurement of serum levels
* Patients must have had a bone marrow biopsy examination in the three months prior to enrolling in the study
* Must be able to provide informed consent
* Systemic and other hematologic causes of pancytopenia, based on clinical presentation, must have been ruled out

Exclusion Criteria:

* Patients with clinically evident congestive heart failure, serious cardiac arrhythmias; symptoms of coronary artery disease must be cleared by cardiology prior to therapy
* Patients who have had chemotherapy, radiotherapy, or immunotherapy or other investigational drug use within 3 weeks prior to study entry
* Pregnant women
* All females of childbearing potential must have a blood test or urine study within two weeks prior to induction registration to rule out pregnancy
* Women of childbearing potential are strongly advised to use an accepted and effective method of contraception
* Patients who have medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Maciejewski, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Afable MG 2nd, Shaik M, Sugimoto Y, Elson P, Clemente M, Makishima H, Sekeres MA, Lichtin A, Advani A, Kalaycio M, Tiu RV, O'Keefe CL, Maciejewski JP. Efficacy of rabbit anti-thymocyte globulin in severe aplastic anemia. Haematologica. 2011 Sep;96(9):1269-75. doi: 10.3324/haematol.2011.042622. Epub 2011 May 23. PMID 21606164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with severe aplastic anemia were recruited over a period of four years (2005-2009) in the hematology clinic at the Cleveland Clinic, a hospital in Cleveland, Ohio.
Groups:
- Rabbit Antithymocyte Globulin (r-ATG/Thymoglobulin): Patients received rabbit anti-thymocyte globulin IV daily over 4-24 hours on days 1-5 (3.5 mg/kg/day). Beginning on day 6, patients received oral cyclosporine twice daily (5 mg/kg/day) for a period of 6 months and then tapered.
Period: Overall Study
Arm/Group | Rabbit Antithymocyte Globulin (r-ATG/Thymoglobulin)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- rATG: Patients receive anti-thymocyte globulin IV daily over 4-24 hours on days 1-5. Beginning on day 6, patients receive oral cyclosporine twice daily for 6 months followed by a taper. Treatment continues in the absence of disease progression or unacceptable toxicity
Arm/Group | rATG
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.95 (18.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Patients Treated With Rabbit Antithymocyte Globulin (r-ATG/Thymoglobulin) and Cyclosporine (CsA) Achieving at Least a Partial Remission (PR) at 6 Months
Description: Patients will be classified as responders if they have transfusion independence and meet two of the following three criteria: ANC greater than 500/mm3; platelet count greater than 20,000/mm3; and reticulocyte count greater than 40,000/mm3. Transfusion independence is defined as no need for transfusions for one month prior to response assessment.
Time Frame: At 6 months
Measure: Number; unit: participants
Arm/Group | Rabbit Antithymocyte Globulin (r-ATG/Thymoglobulin)
Number analyzed (Participants) | 20
participants | 9

ADVERSE EVENTS:
Description: The endpoints of this study evaluated response only. As such, data on non-serious adverse events were not collected or reported for any patients on this trial. Data regarding serious adverse events were collected and reported according to FDA and IRB policies and regulations.
Arm/Group | rATG
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rATG (N=20)
chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
colitis (Infections and infestations) | 2 (2)
compression fractures (Musculoskeletal and connective tissue disorders) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 3 (4)
gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
headache (General disorders) | 1 (1)
pneumonia (Infections and infestations) | 1 (2)
sepsis (Infections and infestations) | 4 (4)
serum sickness (Immune system disorders) | 2 (2)
urinary tract infection (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No